CLINICAL TRIAL: NCT01542086
Title: Comparison of the Cost-Effectiveness of Coronary CT Angiography Versus Myocardial SPECT in Patients With Intermediate Risk of Coronary Heart Disease
Acronym: CARE-CCTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government); Seoul St. Mary's Hospital (Other); Samsung Medical Center (Other); Severance Hospital (Other); Asan Medical Center (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yong-Jin Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-1105-050-361
Record Dates: First submitted 2012-02-14; First posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Chest Pain; Coronary Heart Disease Risk
Keywords: intermediate pre-test; probability of significant coronary heart disease
MeSH Terms: conditions — Chest Pain

ARMS (2):
- Myocardial SPECT (Active Comparator)
  Interventions: Procedure: Myocardial SPECT
- 64-channel coronary CT angiography (CCTA) (Experimental)
  Interventions: Procedure: 64-channel coronary CT angiography (CCTA)

INTERVENTIONS:
Procedure: Myocardial SPECT
  Arms: Myocardial SPECT
Procedure: 64-channel coronary CT angiography (CCTA)
  Arms: 64-channel coronary CT angiography (CCTA)

SUMMARY:
The investigators aim to compare the cost-effectiveness of CCTA and myocardial SPECT in patients with intermediate pre-test probability of CHD. To this end, patients with intermediate pre-test probability of CHD will be randomized 1:1 to either CCTA and myocardial SPECT. The patients will be analyzed for cost and also, for outcome.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the leading cause of heart failure in Westernized countries and accounts for one of the most common cause of mortality in Korea. More importantly, the nation's health cost is being more and more spent on the treatment of CHD. Therefore, selecting the right patients for intervention is becoming more and more important.

The diagnosis and treatment strategy of CHD relies on both anatomic and functional imaging. First, there should be a significant narrowing of a segment of the coronary artery and second, there must also be evidence of ischemia due to the lesion. As a consequence of the recent, rapid development and distribution of the high-resolution computed tomography (CT), physicians are referring more and more patients for anatomic imaging of the coronary vasculature with coronary CT angiography (CCTA). CCTA has the advantage of imaging the coronary arteries noninvasively that is nearly as exact as conventional, invasive coronary angiography. However, CCTA also has the possibility of overdiagnosing CHD, especially intermediate lesions. This can be important give the recent outcome of the FAME study demonstrating the inferiority of relying on only anatomic diagnosis.

In contrast, myocardial single photon emission computed tomography (SPECT) has the advantage of imaging ischemia more accurately, since it is more of a functional imaging than an anatomical imaging. However, the sensitivity and specificity is less than 80%, which means that a total of 20% of the patients can be false-negative or false-positive. In addition, although it can demonstrate ischemia, it cannot provide where and how much the coronary artery is stenotic.

Recently, van Werkhoven and Bax demonstrated that CCTA and myocardial SPECT may be complementary. The study showed that patients with both abnormal CCTA and myocardial SPECT results tend to be worse in terms of event-free survival than patients with either alone. However, the nation's cost may be too burdenful if the patients are charged with both tests together and thus, it is more critical to give information on the cost-effectiveness of both of these tests.

In this study, we aim to compare the cost-effectiveness of CCTA and myocardial SPECT in patients with intermediate pre-test probability of CHD. To this end, patients with intermediate pre-test probability of CHD will be randomized 1:1 to either CCTA and myocardial SPECT. The patients will be analyzed for cost and also, for outcome.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥30 years old and ≤80 years old.
* Subject is able to verbally confirm understandings of risks, benefits and diagnostic alternatives of receiving CCTA or SPECT.
* He/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject must have intermediate probability of coronary artery disease as assessed by the appropriate criteria written below.

Exclusion Criteria:

* The patient has been previously diagnosed as having significant coronary artery disease previously (≥50% stenosis) or has previously been intervened for significant coronary artery disease (PCI or CABG).
* The patient has prior history of myocardial infarction.
* The patient has high pre-test probability of having coronary artery disease.
* The patient has history of impaired renal function, i.e. CRF or ARF.
* The patient has allergy to iodinated contrast agents.
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment), i.e. malignancy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2011-09

PRIMARY OUTCOMES:
Cost-effectiveness (cost-utility) | 1 Year after initial enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea